CLINICAL TRIAL: NCT07394205
Title: Clinical Study of CBG131 CAR-T Cell Injection for the Treatment of CLDN18.2-Positive Advanced Gastric and Pancreatic Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Carbiogene Therapeutics Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2025 No. (005)
Record Dates: First submitted 2026-01-21; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Advanced Gastric and Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBG131 CAR-T Cell Injection (Experimental): This Phase I trial follows a conventional 3 + 3 dose-escalation schema. The dose cohorts are designed as follows: (1) DL1 (de-escalation cohort): 0.5×10⁸ CAR⁺ T cells; (2) DL1 (starting dose cohort): 1×10⁸ CAR⁺ T cells; (3) DL2: 2×10⁸ CAR⁺ T cells. Three subjects are enrolled in each cohort.The dose escalation rule is as follows: Absence of Dose-Limiting Toxicity (DLT) permits escalation to the next higher cohort; one DLT triggers expansion of the current cohort by three additional subjects at the same dose. If one or more additional DLTs occur during the expansion phase: (1) For the DL1 (starting dose cohort), dose escalation is suspended and de-escalation is considered; (2) For DL2 or higher cohorts, dose escalation stops, and the preceding dose is declared as the Maximum Tolerated Dose (MTD). If no further DLTs occur during expansion, dose escalation proceeds.
  Interventions: Drug: CBG131 CAR-T Cell Infusion

INTERVENTIONS:
Drug: CBG131 CAR-T Cell Infusion — This Phase I trial follows a conventional 3 + 3 dose-escalation schema. Cohorts: (1) DL1 (de-escalation cohort): 0.5×10⁸ CAR⁺ T cells; (2) DL1 (starting dose cohort): 1×10⁸ CAR⁺ T cells; (3) DL2: 2×10⁸ CAR⁺ T cells. Three subjects are enrolled in each cohort. Absence of Dose-Limiting Toxicity (DLT) permits dose escalation; one DLT triggers expansion of the cohort by three additional subjects at the same dose. If, during expansion, one or more additional DLTs occur: (1) in the DL1 (starting dose cohort), dose escalation is suspended and de-escalation is considered; (2) in DL2 or higher cohorts, dose escalation stops and the preceding dose is declared the Maximum Tolerated Dose (MTD). If no further DLTs appear, dose escalation proceeds.

SUMMARY:
The goal of this clinical trial is to learn if CBG131 works to treat advanced gastric cancer or pancreatic cancer in adults whose tumors are CLDN18.2-positive. It will also learn about the safety of CBG131 and find the best dose to use.

The main questions it aims to answer are:

Is CBG131 safe, and what medical problems do participants have when receiving it? Does CBG131 shrink tumors in participants with CLDN18.2-positive cancers? How long do the CAR-T cells stay and work in the body? Researchers will test different doses of CBG131 to see which dose is safest and most effective. This is an early-stage trial, so there is no placebo group-everyone who joins will receive the actual treatment.

Participants will:

Have their blood cells collected through a procedure called leukapheresis (so the CAR-T cells can be made).

Receive chemotherapy for 3 days to prepare their body for the CAR-T cells Get a single infusion of CBG131 CAR-T cells through an IV. Visit the clinic frequently for the first month, then regularly for 2 years for checkups, blood tests, and tumor assessments.

Keep track of their symptoms and any side effects they experience.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years (inclusive) at the time of informed consent; sex unrestricted.
2. Voluntary participation: the subject (or legally authorized representative) must provide written informed consent (ICF, Informed Consent Form).
3. Histologically confirmed advanced gastric or gastroesophageal junction adenocarcinoma that has progressed after ≥ 2 prior systemic regimens, OR histologically confirmed advanced pancreatic adenocarcinoma that has progressed after ≥ 1 prior systemic regimen.
4. CLDN18.2 positivity in archival or fresh tumor tissue by immunohistochemistry (IHC): ≥ 40% of tumor cells staining ≥ 2+.
5. At least one measurable lesion per RECIST 1.1 (longest diameter ≥ 10 mm).
6. Estimated life expectancy > 12 weeks.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
8. Adequate organ function within 14 days prior to leukapheresis, defined by all of the following:

(1) Total bilirubin ≤ 2 × ULN (Upper Limit of Normal); (2) ALT and AST ≤ 2.5 × ULN (≤ 5 × ULN if liver or bone metastases are present); (3) Calculated creatinine clearance (Cockcroft-Gault) ≥ 50 mL/min; (4) Hemoglobin ≥ 90 g/L; (5) White blood cell (WBC) count ≥ 1.5 × 10⁹/L, with documented suitable venous access for leukapheresis and no contraindications to leukapheresis; (6) Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L without Granulocyte Colony-Stimulating Factor (G-CSF) or other myeloid growth factors within 7 days of screening labs; (7) Absolute lymphocyte count ≥ 0.5 × 10⁹/L; (8) Platelet count ≥ 80 × 10⁹/L without transfusion within 7 days of screening labs; (9) Prothrombin time (PT) prolongation ≤ 4 s above ULN; (10) Oxygen saturation ≥ 95% on room air. 9: Contraception and pregnancy requirements: Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and again before lymphodepleting chemotherapy; must not be breastfeeding. WOCBP and fertile men must use a highly effective contraceptive method from screening until 12 months after CBG131 infusion or study discontinuation, whichever is later.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Active bacterial or fungal infection within 72 h before lymphodepletion. Subjects receiving prophylactic antibiotics, antifungals or antivirals are allowed if there is no evidence of active infection and the agents are not on the prohibited-medication list.
3. Systemic corticosteroids equivalent to > 15 mg/day prednisone within 2 weeks before leukapheresis (inhaled or topical steroids permitted). Any systemic glucocorticoids within 7 days before leukapheresis, except inhaled or topical preparations.
4. Live-attenuated vaccine within 4 weeks before leukapheresis or planned during the study.
5. Positive HBsAg or HBcAb with HBV-DNA ≥ ULN; positive HCV antibody with detectable HCV RNA; positive HIV antibody; positive syphilis serology.
6. Prior hypersensitivity to immunotherapy, cyclophosphamide, fludarabine, albumin-bound paclitaxel, tocilizumab, or any component of CBG131 (e.g. DMSO), or other significant allergic history.
7. Anti-cancer therapy within 2 weeks before leukapheresis (or 5 half-lives, whichever is shorter), including surgery, systemic chemotherapy, radiotherapy, interventional procedures, or anti-PD-1/PD-L1 monoclonal antibody (mAb)/Claudin18.2-targeted agents/other investigational drugs within 4 weeks (or 5 half-lives).
8. Prior gene-engineered cellular therapy (e.g. CAR-T, TCR-T, TIL).
9. Major surgery within 4 weeks before leukapheresis or significant trauma, or anticipated major surgery during the study (except cataract or local-anaesthetic procedures).
10. Known or suspected brain metastases.
11. Portal-vein tumor thrombus or tumor thrombus in mesenteric/inferior vena cava on imaging.
12. Central or extensive pulmonary metastases, extensive liver metastases, or widespread bone metastases.
13. History of organ transplantation or on transplant waiting list.
14. Uncontrolled or serious illnesses that could limit participation, including: Diabetes with HbA1c > 8%, uncontrolled hypertension (> 160/100 mmHg), Left Ventricular Ejection Fraction (LVEF) < 50%, congestive heart failure, acute MI, severe arrhythmia, unstable angina within 6 months, pulmonary embolism, COPD, ILD, clinically significant pulmonary-function abnormalities; Active peptic ulcer, active GI bleeding, bleeding diathesis, major GI bleed within 3 months, prior immunotherapy-related bleeding, hypotension requiring vasopressors.
15. Deep ulceration of primary tumor, full-thickness infiltration at anastomotic recurrence, or tumor encasing/invading major vessels on CT/MRI ± endoscopy, carrying high risk of bleeding or perforation.
16. Requirement for warfarin or heparin anticoagulation.
17. Chronic antiplatelet therapy at doses exceeding aspirin 100 mg/day or clopidogrel 75 mg/day.
18. Toxicities from prior therapies not resolved to ≤ Grade 1 or baseline (except alopecia, pigmentation, or laboratory abnormalities allowed by protocol) at informed-consent signature.
19. Clinically significant CNS disease, abnormal neurologic findings, or psychiatric disorder.
20. Other malignancies within 5 years (except adequately treated cervical carcinoma in situ or basal-cell skin cancer).
21. Clinically relevant thyroid dysfunction (TT4, TT3, FT3, FT4, TSH outside normal limits per investigator).
22. Active autoimmune disease (e.g. psoriasis, RA) or any condition requiring chronic immunosuppressive therapy.
23. Known or suspected CNS metastases.
24. Single target lesion > 4 cm in longest diameter (or > 4 cm short axis for lymph nodes) before leukapheresis.
25. Symptomatic ascites or ascites requiring repeated paracentesis or intraperitoneal therapy; small-volume radiologic ascites permitted if asymptomatic.
26. Any other condition that, in the opinion of the investigator, renders the subject unsuitable for participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-09-30 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and Grading of Adverse Events (AEs) and Serious Adverse Events (SAEs)（Including CRS and ICANS） | From leukapheresis enrollment up to 15 years post-CBG131 infusion, or until study withdrawal, loss to follow-up, or death of the subject, whichever comes first.
  This outcome measure assesses the incidence and severity grading of all Adverse Events (AEs) and Serious Adverse Events (SAEs) in subjects. Specifically: a) Cytokine Release Syndrome (CRS) and Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) are graded according to the ASTCT (American Society for Transplantation and Cellular Therapy) consensus criteria; b) All other AEs are graded according to the NCI-CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) Version 5.0. Data are collected from leukapheresis enrollment to the end of the follow-up period.
Incidence and Determination of Dose-Limiting Toxicity (DLT) Related to CBG131 | Within 28 days after CAR-T cell infusion.
  Dose-Limiting Toxicity (DLT) refers to CBG131-related toxicities (excluding infections and malignancies) occurring within 28 days after CAR-T cell infusion. DLT is determined based on the following criteria: 1) Grade 5 AE; 2) Grade 4 CRS; 3) Grade 4 neurotoxicity; 4) Grade 3 CRS or neurotoxicity that persists for more than 72 hours and fails to improve to ≤Grade 2; 5) Other Grade 4 non-hematologic toxicity that persists for more than 72 hours and fails to improve to ≤Grade 3; 6) Other Grade 3 non-hematologic toxicity that persists for ≥2 weeks; 7) Grade 4 hematologic toxicity that persists for more than 72 hours and fails to improve to ≤Grade 3; 8) Hematologic toxicity of Grade >3 that persists for more than 2 weeks and fails to improve to ≤Grade 2.
Maximum Tolerated Dose (MTD) and Optimal Dosage of CBG131（Determined by 3+3 Dose-Escalation Schema） | Within 28 days after CAR-T cell infusion (DLT assessment period); the MTD is determined after completion of dose escalation for all cohorts.
  This Phase I trial adopts a conventional 3 + 3 dose-escalation schema to determine the Maximum Tolerated Dose (MTD) of CBG131 and further confirm its optimal dosage. The dose cohorts are designed as follows: (1) DL1 (de-escalation cohort): 0.5×10⁸ CAR⁺ T cells; (2) DL1 (starting dose cohort): 1×10⁸ CAR⁺ T cells; (3) DL2: 2×10⁸ CAR⁺ T cells. Three subjects are enrolled in each cohort. If no DLT occurs in a cohort, dose escalation proceeds to the next higher cohort; if one DLT occurs, the cohort is expanded by an additional three subjects at the same dose. During the expansion phase: (1) If one or more additional DLTs occur in the DL1 (starting dose cohort), dose escalation is suspended and de-escalation is considered; (2) If one or more additional DLTs occur in DL2 or higher cohorts, dose escalation stops, and the previous dose is declared as the MTD. If no additional DLTs occur during expansion, dose escalation continues.

SECONDARY OUTCOMES:
Tumor CLDN18.2 Expression Positivity (Assessed by Immunohistochemistry [IHC]) | Screening period (before CAR-T cell infusion).
  This outcome measure assesses the positivity of CLDN18.2 expression in primary tumor tissue of subjects. Primary tumor tissue samples obtained within ≤1 year after subject consent must be detected for CLDN18.2 expression by Immunohistochemistry (IHC), and the expression positivity is determined according to the predefined IHC criteria.
Progression-Free Survival (PFS) per RECIST 1.1 Criteria | From the date of CBG131 infusion to the first documented evidence of disease progression or death from any cause, whichever occurs first; assessed up to Week 48 (±7 days), with interim assessments at Weeks 6, 12, 18, 24, 36 and 48 (±7 days).
  Progression-Free Survival (PFS) is defined and calculated according to the RECIST (Response Evaluation Criteria in Solid Tumors) Version 1.1 for efficacy evaluation. PFS refers to the interval from the date of CBG131 infusion to the first documented evidence of disease progression or death from any cause, whichever occurs first. Disease progression is determined in accordance with RECIST 1.1 criteria.
Overall Survival (OS) | From the date of CBG131 infusion to death from any cause, whichever occurs first; assessed up to 2 years post-treatment (or until loss to follow-up, withdrawal of consent, or death, whichever comes first), with follow-up every 3 months (±2 weeks).
  Overall Survival (OS) is defined as the interval from the date of CBG131 infusion to death from any cause. After CAR-T cell infusion, all subjects who discontinue the study for any reason will undergo survival follow-up every 3 months (±2 weeks) until the end of the follow-up period.
Best Overall Response Rate (BORR) per RECIST 1.1 Criteria（Proportion of Subjects Achieving Complete Response [CR] or Partial Response [PR]） | Weeks 6, 12, 18, 24, 36 and 48 (±7 days); the best overall response of each subject is determined based on the responses recorded at all above time points.
  The Best Overall Response Rate (BORR) is evaluated according to the RECIST 1.1 criteria for antitumor response. Antitumor responses are classified into four categories: Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD). BORR is defined as the proportion of subjects who achieve CR or PR during the study period. The number and percentage of subjects achieving CR or PR will be tabulated, and the 95% confidence interval for each percentage will be calculated using the Clopper-Pearson exact method. For the calculation of BORR, each subject's best response recorded at any time during the study will be used.
CAR-T Cell Persistence in Vivo (Assessed by Peripheral Blood qPCR for CAR Transgene Copies [copies/μg gDNA]) | Assessed at Day 1, Day 4, Day 7, Day 11, Day 15, Day 21;Week 4, Week 6, Week 12, Week 18, Week 24, Week 36, Week 48;every 6 Months(±2 Months) during Years 2 to 5;every 12 Months(±2 Months) during Years 5 to 15;assessed up to 15 years post-CBG131 infusion
  This outcome measure assesses the persistence of CAR-T cells in the peripheral blood of subjects in vivo. Peripheral blood samples are collected at predefined time points, and the number of CAR transgene copies in the samples is detected by quantitative Polymerase Chain Reaction (qPCR) with the unit of copies/μg gDNA. The persistence of CAR-T cells is evaluated based on the dynamic changes of CAR transgene copy number over time.
Serum Interleukin-2 (IL-2) Concentration (Assessed by Lab Cytokine Assay) | Baseline, Day 0, Day 1, Day 4, Day 7, Day 11, Day 15, Day 21, Week 4, Week 6.
  This outcome measure assesses the concentration of Interleukin-2 (IL-2) in the serum of subjects. Serum samples are collected at predefined time points, and IL-2 concentration is detected by standard lab cytokine assays. IL-2 is a cytokine involved in immune regulation, and its concentration change reflects the immune response status of subjects after treatment.
3-month Objective Response Rate (ORR) per RECIST 1.1 Criteria（Proportion of Subjects Achieving CR or PR） | Within 3 months (±7 days) after CBG131 infusion.
  The 3-month Objective Response Rate (ORR) is evaluated according to the RECIST 1.1 criteria. It is defined as the proportion of subjects who achieve Complete Response (CR) or Partial Response (PR) within 3 months after CBG131 infusion. The response status of subjects is determined by tumor assessment according to RECIST 1.1 criteria at the 3-month time point.
Duration of Response (DOR) per RECIST 1.1 Criteria | From the date of first documented CR or PR to the date of first documented disease progression (per RECIST 1.1 criteria) or death from any cause, whichever occurs first; assessed up to 15 years post-CBG131 infusion.
  Duration of Response (DOR) is defined as the interval from the date of first documented Complete Response (CR) or Partial Response (PR) to the date of first documented evidence of disease progression (assessed by RECIST 1.1 criteria) or death from any cause, whichever occurs first. This outcome measure is only applicable to subjects who achieve an objective response (CR or PR) after CBG131 infusion.
Time to Response (TTR) per RECIST 1.1 Criteria | From the date of CBG131 infusion to the first documented CR or PR; assessed up to Week 48 (±7 days) (if no response is documented by Week 48, TTR is considered not achieved).
  Time to Response (TTR) is defined as the interval from the date of CBG131 infusion to the date of first documented objective response (including CR and PR) in subjects who achieve an objective response. TTR is described using statistical indicators including mean, median, standard deviation, minimum, and maximum. If no objective response is documented by Week 48 post-infusion, TTR is considered not achieved.
Duration of Disease Control (DDC) per RECIST 1.1 Criteria | From the date of first documented CR, PR, or SD (per RECIST 1.1 criteria) to the date of first documented PD or death from any cause, whichever occurs first; assessed up to 15 years post-CBG131 infusion.
  Duration of Disease Control (DDC) is defined as the interval from the date of first documented Complete Response (CR), Partial Response (PR), or Stable Disease (SD) to the date of first documented Progressive Disease (PD) or death from any cause, whichever occurs first. DDC reflects the duration of disease control in subjects after treatment, and it will be statistically described using mean, median, standard deviation, minimum, and maximum.
Correlation Between Tumor CLDN18.2 Expression Level (Assessed by IHC) and Efficacy Endpoints (Post-hoc Analysis) | Post-hoc correlation analysis between tumor CLDN18.2 level and efficacy endpoints; analysis will be performed after completion of efficacy follow-up (assessed up to 15 years post-CBG131 infusion).
  This outcome measure is a post-hoc analysis to explore the correlation between tumor CLDN18.2 expression level (assessed by IHC) and efficacy endpoints (including PFS, OS, ORR, DOR, etc.). Logistic regression and Cox proportional hazards regression models are used for statistical analysis. An exploratory cut-off value of H-score ≥200 is adopted to classify the CLDN18.2 expression level, and the correlation between different expression levels and efficacy endpoints is analyzed.
Serum Soluble PD-L1 Concentration（Central Lab） | Screening, Baseline, Week 6, Week 12, Week 18, Week 24, Week 36, Week 48.
  This outcome measure assesses the concentration of soluble programmed death-ligand 1 (sPD-L1) in the serum of subjects. Serum samples are collected at predefined time points, and soluble PD-L1 concentration is detected by the central laboratory using standard lab assays.
Serum CA125 Level（Site Lab） | Screening, Baseline, Week 6, Week 12, Week 18, Week 24, Week 36, Week 48.
  This outcome measure assesses the level of carbohydrate antigen 125 (CA125) in the serum of subjects. Serum samples are collected at predefined time points, and CA125 level is detected by the site laboratory using standard lab assays. CA125 is a tumor marker used for auxiliary assessment of disease status.
Serum Carcinoembryonic Antigen (CEA) Level（Site Lab） | Screening, Baseline, Week 6, Week 12, Week 18, Week 24, Week 36, Week 48.
  This outcome measure assesses the level of carcinoembryonic antigen (CEA) in the serum of subjects. Serum samples are collected at predefined time points, and CEA level is detected by the site laboratory using standard lab assays. CEA is a tumor marker used for auxiliary assessment of disease status.
Serum Carbohydrate Antigen 19-9 (CA19-9) Level（Site Lab） | Screening, Baseline, Week 6, Week 12, Week 18, Week 24, Week 36, Week 48.
  This outcome measure assesses the level of carbohydrate antigen 19-9 (CA19-9) in the serum of subjects. Serum samples are collected at predefined time points, and CA19-9 level is detected by the site laboratory using standard lab assays. CA19-9 is a tumor marker used for auxiliary assessment of disease status.
CAR-T Cell Peak Expansion in Vivo (Assessed by Peripheral Blood qPCR for CAR Transgene Copies [copies/μg gDNA]) | Assessed at Day 1, 4, 7, 11, 15, 21; Week 4, 6, 12, 18, 24, 36, 48; every 6 Months (±2 Months) in Years 2-5; every 12 Months (±2 Months) in Years 5-15; peak expansion determined up to 15 years post-infusion.
  This outcome measure assesses the peak expansion level of CAR-T cells in the peripheral blood of subjects in vivo. Peripheral blood samples are collected at predefined time points, and the number of CAR transgene copies in the samples is detected by qPCR with the unit of copies/μg gDNA. The peak expansion level is defined as the maximum value of CAR transgene copy number detected during the follow-up period.
Area Under the Curve (AUC) of CAR-T Cell Expansion in Vivo (Assessed by Peripheral Blood qPCR for CAR Transgene Copies [copies/μg gDNA]) | Assessed at Days 1,4,7,11,15,21; Weeks 4,6,12,18,24,36,48; every 6 Months (±2 Months) during Years 2 to 5; every 12 Months (±2 Months) during Years 5 to 15; AUC is calculated based on all detected data up to 15 years post-CBG131 infusion.
  This outcome measure assesses the Area Under the Curve (AUC) of CAR-T cell expansion in the peripheral blood of subjects in vivo, which reflects the overall expansion level of CAR-T cells during the follow-up period. Peripheral blood samples are collected at predefined time points, and the number of CAR transgene copies is detected by qPCR. The AUC is calculated based on the dynamic curve of CAR transgene copy number over time, with the unit of copies/μg gDNA × time.
Serum Interleukin-6 (IL-6) Concentration (Assessed by Lab Cytokine Assay) | Baseline, Day 0, Day 1, Day 4, Day 7, Day 11, Day 15, Day 21, Week 4, Week 6.
  This outcome measure assesses the concentration of Interleukin-6 (IL-6) in the serum of subjects. Serum samples are collected at predefined time points, and IL-6 concentration is detected by standard lab cytokine assays. IL-6 is a cytokine closely related to CRS, and its concentration change is used for auxiliary assessment of CRS severity.
Serum Interferon-γ (IFN-γ) Concentration (Assessed by Lab Cytokine Assay) | Baseline, Day 0, Day 1, Day 4, Day 7, Day 11, Day 15, Day 21, Week 4, Week 6.
  This outcome measure assesses the concentration of Interferon-γ (IFN-γ) in the serum of subjects. Serum samples are collected at predefined time points, and IFN-γ concentration is detected by standard lab cytokine assays. IFN-γ is an immune-regulatory cytokine that reflects the anti-tumor immune response of subjects.
Serum Tumor Necrosis Factor-α (TNF-α) Concentration (Assessed by Lab Cytokine Assay) | Baseline, Day 0, Day 1, Day 4, Day 7, Day 11, Day 15, Day 21, Week 4, Week 6.
  This outcome measure assesses the concentration of Tumor Necrosis Factor-α (TNF-α) in the serum of subjects. Serum samples are collected at predefined time points, and TNF-α concentration is detected by standard lab cytokine assays. TNF-α is a pro-inflammatory cytokine involved in the immune response and inflammation regulation after treatment.
Serum C-X-C Motif Chemokine Ligand 10 (CXCL10) Concentration (Assessed by Lab Cytokine Assay) | Baseline, Day 0, Day 1, Day 4, Day 7, Day 11, Day 15, Day 21, Week 4, Week 6.
  This outcome measure assesses the concentration of C-X-C Motif Chemokine Ligand 10 (CXCL10) in the serum of subjects. Serum samples are collected at predefined time points, and CXCL10 concentration is detected by standard lab cytokine assays. CXCL10 is a chemokine involved in immune cell recruitment and anti-tumor immune response.
Serum Interleukin-8 (IL-8) Concentration (Assessed by Lab Cytokine Assay) | Baseline, Day 0, Day 1, Day 4, Day 7, Day 11, Day 15, Day 21, Week 4, Week 6.
  This outcome measure assesses the concentration of Interleukin-8 (IL-8) in the serum of subjects. Serum samples are collected at predefined time points, and IL-8 concentration is detected by standard lab cytokine assays. IL-8 is a pro-inflammatory chemokine involved in neutrophil recruitment and inflammation response after treatment.
Serum Monocyte Chemoattractant Protein-1 (MCP-1) Concentration (Assessed by Lab Cytokine Assay) | Baseline, Day 0, Day 1, Day 4, Day 7, Day 11, Day 15, Day 21, Week 4, Week 6.
  This outcome measure assesses the concentration of Monocyte Chemoattractant Protein-1 (MCP-1) in the serum of subjects. Serum samples are collected at predefined time points, and MCP-1 concentration is detected by standard lab cytokine assays. MCP-1 is a chemokine that mediates monocyte recruitment and participates in immune regulation and inflammation response.
Serum Interferon-α2 (IFN-α2) Concentration (Assessed by Lab Cytokine Assay) | Baseline, Day 0, Day 1, Day 4, Day 7, Day 11, Day 15, Day 21, Week 4, Week 6.
  This outcome measure assesses the concentration of Interferon-α2 (IFN-α2) in the serum of subjects. Serum samples are collected at predefined time points, and IFN-α2 concentration is detected by standard lab cytokine assays. IFN-α2 is an antiviral and immune-regulatory cytokine that participates in the anti-tumor immune response of subjects.
Serum TGF-β1 Concentration（Central Lab） | Screening, Baseline, Week 6, Week 12, Week 18, Week 24, Week 36, Week 48.
  This outcome measure assesses the concentration of transforming growth factor-β1 (TGF-β1) in the serum of subjects. Serum samples are collected at predefined time points, and TGF-β1 concentration is detected by the central laboratory using standard lab assays.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, study protocol and metadata will be made publicly available within 6 months after study completion on the ClinicalTrials.gov at https://clinicaltrials.gov.